CLINICAL TRIAL: NCT00982982
Title: Gamma-Amino Butyric Acid (GABA) Deficits and Vulnerability to Cannabinoid-Induced Psychosis
Brief Title: Effects of Delta-9-THC and Iomazenil in Healthy Humans
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Associate Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 0901004662
Record Dates: First submitted 2009-08-18; First posted 2009-09-23 (Estimated); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Schizophrenia; Mental Disorders; Psychotic Disorders
Keywords: Schizophrenia; Mental Disorders; Psychotic Disorders; Schizophrenia and Disorders with Psychotic Features; Cannabis
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Psychotic Disorders; Schizophrenia Spectrum and Other Psychotic Disorders; Marijuana Abuse | interventions — Dronabinol; iomazenil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- THC and Iomazenil (Active Comparator): * Iomazenil: 3.7 μg/kg intravenously over 10 minutes
  * Delta-9-THC (0.015 mg/kg = 1.05 mg in a 70kg individual), dissolved in alcohol. This dose is roughly equivalent to smoking approximately 1/4th of a marijuana cigarette, or "joint". It is administered intravenously for 10 minutes
  Interventions: Drug: THC and Iomazenil
- Placebo (Placebo Comparator): Control: small amount of alcohol intravenous (quarter teaspoon), with no THC
  Interventions: Drug: Placebo (control)

INTERVENTIONS:
Drug: THC and Iomazenil — * Iomazenil: 3.7 μg/kg intravenously over 10 minutes
  * Delta-9-THC (0.015 mg/kg = 1.05 mg in a 70kg individual), dissolved in alcohol. This dose is roughly equivalent to smoking approximately 1/4th of a marijuana cigarette, or "joint". It is administered intravenously for 10 minutes.
  Arms: THC and Iomazenil
Drug: Placebo (control) — Control: small amount of alcohol intravenous (quarter teaspoon), with no THC
  Arms: Placebo

SUMMARY:
The study aims to examine the combined effects of delta-9-tetrahydrocannabinol (∆-9-THC or THC) and iomazenil on thinking, perception, mood, memory, attention, and electrical activity of the brain (EEG). THC is the active ingredient of marijuana, cannabis, "ganja", or "pot". Iomazenil is a drug that works opposite to drugs like valium. The purpose of this study is to determine whether the administration of iomazenil will alter the effects of THC.

ELIGIBILITY:
Inclusion Criteria:

* Exposed to cannabis at least once in their lifetime

Exclusion Criteria:

* Cannabis naïve
* History of hearing deficit

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2009-02-11 (Actual); Primary Completion 2013-02-22 (Actual); Study Completion 2013-02-22 (Actual)

PRIMARY OUTCOMES:
Clinician Administered Dissociative Symptoms Scale | On each test day at: baseline, +10min after infusion, +70min, +150min, +240min
Positive and Negative Symptom Scale | On each test day at: baseline, +10min after infusion, +70min, +150min, +240min
Visual Analog Scale | On each test day at: baseline, +10min after infusion, +70min, +150min, +240min
Auditory Verbal Learning Test | On each test day at: baseline, +10min after infusion, +70min, +150min, +240min
Perceptual Aberration Scale | On each test day at: baseline, +10min after infusion, +70min, +150min, +240min

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C D'Souza, M.D, Principal Investigator — Yale University Medical School
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States